CLINICAL TRIAL: NCT00874978
Title: The Efficacy and Safety of Lenalidomide (Revlimid®) Monotherapy in Red Blood Cell Transfusion Dependent Subjects With Myelodysplastic Syndrome Associated With Del (5q) Cytogenetic Abnormality
Brief Title: The Efficacy and Safety of Lenalidomide Monotherapy in Red Blood Cell Transfusion Dependent Subjects With Myelodysplastic Syndrome (MDS) Associated With Del (5q) Abnormality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Professor Ghulam Mufti, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04CC06; REC - 04/Q0703/148; EudraCT - 2004-005101-29
Record Dates: First submitted 2009-03-16; First posted 2009-04-03 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2015-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Lenalidomide; myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Oral lenalidomide 10mg (two 5mg capsules) daily on days 1-21 every 28 days for up to 6 cycles.
  Other Names: Revlimid; CC-5013

SUMMARY:
The purpose of this study is to evaluate the efficacy of lenalidomide treatments to achieve haematopoietic improvement in subjects with low- or intermediate-1 risk International Prognostic Scoring System1 (IPSS) myelodysplastic syndrome (MDS) associated with a del (5q31-33) cytogenetic abnormality.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age over or equal to 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosis of low- or intermediate-1-risk (IPSS) MDS associated with a del(5q) cytogenetic abnormality. The cytogenetic abnormality of chromosome 5 must involve a deletion between bands q31 and q33. The del(5q) cytogenetic abnormality may be an isolated finding or may be associated with other cytogenetic abnormalities.
5. RBC transfusion-dependent anaemia defined as having no transfusion free interval of < 56 consecutive days within the past 112 days.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
7. Women of childbearing potential (WCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study drug and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. Women must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.
8. Laboratory test results within these ranges:

   * Absolute neutrophil count over or equal to 0.5 x 109/L
   * Platelet count over or equal to 25 x 109/L
   * Serum creatinine under or equal to 2.0 mg/dl
   * Total bilirubin under or equal to 1.5 mg/dl
   * AST (SGOT) and ALT (SGPT) under or equal to 3 x ULN.
9. Disease free of prior malignancies for over or equal to 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Prior > grade 3 (National Cancer Institute [NCI] Common Toxicity Criteria [CTC]) allergic reaction to thalidomide.
4. Prior > grade 3 (NCI CTC) rash or any desquamation (blistering) while taking thalidomide.
5. Clinically significant anaemia due to factors such as iron, B12 or folate deficiencies,autoimmune or hereditary haemolysis or gastrointestinal bleeding (if a marrow aspirate is not evaluable for storage iron, transferrin saturation must be > 20 % and serum ferritin not less than 50 ng/ml).
6. Use of haematopoietic growth factors within 7 days of the first day of study drug treatment. Use of G-CSF is permitted.
7. Concurrent use of erythropoietin
8. Chronic use (>2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to >10 mg/day of prednisolone) within 28 days of the first day of study lenalidomide treatment.
9. Use of experimental or standard drugs (i.e. chemotherapeutic, immunosuppressive, and cytoprotective agents) for the treatment of MDS within 28 days of the first day of study lenalidomide treatment.
10. Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for >3 years.
11. Any prior use of lenalidomide.
12. Concurrent use of other anti-cancer agents or treatments. Patients must not have received any form of chemotherapy for at least 4 weeks prior to study entry and must have fully recovered from haematological toxicity associated with this therapy.
13. Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Red blood cell (RBC) transfusion independence. | monthly

SECONDARY OUTCOMES:
Cytogenetic response | 3, 6 and 12 months
Over or equal to 50% decrease in RBC transfusion requirements | monthly
Change of haemoglobin concentration from baseline | every 2 and 4 weeks
Safety (type, frequency, severity, and relationship of adverse events to lenalidomide) | monthly
Platelet response | every 2 and 4 weeks
Neutrophil response | every 2 and 4 weeks
Bone marrow response | 3, 6 and 12 months
Duration of response | monthly
Gene expression profiling of patients with the 5q- syndrome and effects of lenalidomide on gene expression profiles | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam J Mufti, MB, DM, FRCP, FRCPath, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom